CLINICAL TRIAL: NCT06095349
Title: Effect of Sulfur Thermal Water on Circulating H2S Levels and Markers of Bone Metabolism in Osteopenic Subjects.
Acronym: FORST3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FORST3
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Hydrogen Sulfide; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone turnover markers (Experimental): Concentrations of bone turnover markers will be assessed before and after treatment. Correlation will be sought for with H2S levels and clinical features of the patients
  Interventions: Other: inhalatory treatment with sulfureous aerosol

INTERVENTIONS:
Other: inhalatory treatment with sulfureous aerosol — osteopenic patients are subject to a 12-days cycle of 30 minutes-long inhalatory treatment with sulfureous aerosol

SUMMARY:
The aim of the study is to investigate whether inhalation treatment with high-sulfide waters from some spas (referred to as "thermal waters"), performed for 12 consecutive days, is able to change circulating H2S levels and alter bone metabolism. Identifying a clear correlation between circulating levels of H2S and sulfur water administration, as well as a potential anabolic effect on bone, would set the stage for new studies that could have important clinical implications for promoting health and preventing osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women with a diagnosis of osteopenia

Exclusion Criteria:

* concurrent muscoloskeletal conditions or chronic pharmacological treatment interfering with bone metabolism

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — post-menopausal women, a condition which is associated with the development of osteoporosis
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Measurement of biomarkers of bone turnover, marker #1 | 15 days
  Procollagen type 1 N-terminal propeptide (P1NP), marker of bone formation
Measurement of biomarkers of bone turnover, marker #2 | 15 days
  Bone-specific alkaline phosphatase (BAP), marker of bone formation
Measurement of biomarkers of bone turnover, marker #3 | 15 days
  serum C-terminal telopeptide of type I collagen (CTX-1), marker of bone resorption

SECONDARY OUTCOMES:
Measurement of serum H2S levels | 15 days
  serum H2S levels will be assessed through HPLC

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy